CLINICAL TRIAL: NCT01890837
Title: Effect of Daikenchuto (TU-100), a Gastrointestinal Nerve Modulator, on Rectal Sensation in Patients With Irritable Bowel Syndrome
Brief Title: Effect of TU-100 in Patients With Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tsumura USA (Industry)
Collaborators: Cato Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TU100CPT5
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Irritable Bowel Syndrome; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Abdominal Pain
Keywords: Rectal Compliance; Rectal Sensation; Rectal Tone
MeSH Terms: conditions — Irritable Bowel Syndrome; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Abdominal Pain | interventions — dai-kenchu-to; 12,13-dihydro-N-methyl-6,11,13-trioxo-5H-benzo(4,5)cyclohepta(1,2-b)naphthalen-5,12-imine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daikenchuto (TU-100) 15g/day (Experimental): Daikenchuto (TU-100) 5g TID/3 times per day (15g/day)
  Interventions: Drug: Daikenchuto (TU-100)
- Placebo (Placebo Comparator): Placebo TID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Daikenchuto (TU-100) — Subjects will receive 5g TID (15g/day) of TU-100. Dosage form is granule. Subject will take a daily dose divided 3 times per day for 2 weeks.
  Arms: Daikenchuto (TU-100) 15g/day
Drug: Placebo — Subjects will receive daily dose of TU-100 placebo. Dosage form is granule. Subject will take a daily dose divided 3 times per day for 2 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effects of 5g of Daikenchuto (TU-100) three times per day (Daikenchuto [TU-100] is a botanical agent that modulates gastrointestinal nerves), and placebo on rectal sensation (sensation ratings of urgency to defecate and sensation threshold for pain) in response to rectal balloon distension by barostat in patients with IBS.

ELIGIBILITY:
Inclusion Criteria:

1. Meet Rome III criteria for IBS.
2. Willing and able to provide written informed consent.
3. If a female of childbearing potential, must be using an acceptable form of contraception during the study and for 30 days after the last dose. Acceptable methods include surgical sterilization, hormonal contraceptives (such as oral contraceptives, Depo-Provera, NuvaRing), condoms used with a spermicide, an IUD [Intrauterine device] or abstinence.

   Females are not considered to be of childbearing potential if they are postmenopausal for at least 2 years or have been surgically sterilized.
4. Aged 18 to 65 years, inclusive.
5. Have a body mass index (BMI) between 18 and 40 kg/m2, inclusive.
6. Have a negative urine drug screening at Visit 1.
7. Have normal or not clinically significant laboratory results as reviewed by the study physicians.
8. Have a normal rectal examination result on file within the past 2 years or performed at Visit 1 in order to exclude the possibility of an evacuation disorder (examination must exclude findings suggestive of an evacuation disorder such as high sphincter tone at rest, failure of perineal descent and spasm, tenderness or paradoxical contraction of the puborectalis muscles).
9. Agree to avoid alcohol during the entire study to avoid corrupting the data from the rectal barostat tests.

Exclusion Criteria:

1. Have a structural or metabolic diseases or conditions that affect the GI system.
2. Be taking any medication that in the opinion of the principal investigator has a potential to alter GI transit (this includes but is not limited to osmotic or stimulant laxatives, magnesium or aluminum-containing antacids, prokinetics, erythromycin, gabapentin, pregabalin, narcotics, anticholinergics, antidepressants [including selective norepinephrine reuptake inhibitors], antipsychotics, opiates, GABAergic agents and benzodiazepines).

   Note: Tricyclic antidepressants are permissible at doses equal to or less than 25 mg daily; selective serotonin reuptake inhibitor antidepressants are permissible at low, stable doses. Analgesics such as Tylenol, ibuprofen, naproxen and aspirin are not permissible during Visits 2 and 3 to avoid corrupting data from the rectal barostat tests. All medications will be reviewed by the principal investigator on a case by case basis.

   Rescue medications: Rescue medications will be reviewed and approved as necessary for exacerbation of constipation or diarrhea since the study medication treatment period is about 14 days total. The patient will contact the study staff to request review and approval of the use of a rescue medication by the principal investigator. The use of the rescue medication will be documented by the patient in the bowel pattern, bloating and pain diary. Rescue medications are not allowed within 7 days of the rectal sensation studies to ensure data integrity.
3. Have clinical evidence, including but not limited to, of a clinically significant abnormal physical examination or laboratory value or of a past event documented in the past medical record, or current clinically significant abnormal physical examination or laboratory value that could indicate significant cardiovascular, respiratory, renal, hepatic, GI, hematological, neurological, psychiatric or other diseases that interfere with the objectives of the study. If a laboratory test value falls outside of the reference range and is considered clinically significant, it may be repeated once at the discretion of the principal investigator. If the laboratory test result remains abnormal and clinically significant, the patient will be discontinued from the study and referred to a primary care physician for evaluation.
4. Be a known substance abuser or be considered to be an alcoholic not in remission.
5. Have participated in another clinical study in the past 30 days.
6. Have a history of allergic reactions to egg, ginseng, ginger or Sichuan pepper.
7. Be clinically lactose intolerant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Sensation rating of urgency to defecate in response to 32 mmHg distension of rectum on a 100 mm VAS | 14 days
Sensation threshold for pain in response to distention of the rectum | 14 days

SECONDARY OUTCOMES:
Rectal compliance at half-maximum pressure (Pr1/2) | 14 days
Rectal sensation thresholds (gas, urgency to defecate, first sensation) | 14 days
Rectal sensation ratings (pain, gas) in response to 32 mmHg distension of the rectum | 14 days
Rectal tone response to feeding 1,000 kcal meal | 14 days
Stool frequency | 21 days
Stool consistency as measured by the Bristol stool scale | 21 days
Daily average severity of abdominal pain on 100mm VAS | 21 days
Worst severity of abdominal pain each day measured on 100mm VAS scale | 21 days
Daily average severity of bloating on 100mm VAS scale | 21 days
IBS-QOL (Quality of Life) score | 14 days
Ease of bowel movements | 21 days
Completeness of evacuation | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester Methodist CRU, Rochester, Minnesota, United States